CLINICAL TRIAL: NCT01704716
Title: High Risk Neuroblastoma Study 1 of SIOP-Europe (SIOPEN)
Brief Title: High Risk Neuroblastoma Study 1.8 of SIOP-Europe (SIOPEN)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Anna Kinderkrebsforschung (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-NBL-1.8 / SIOPEN
Record Dates: First submitted 2012-10-05; First posted 2012-10-11 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma; immunotherapy; MAT; antibody treatment
MeSH Terms: conditions — Neuroblastoma | interventions — Vincristine; aldesleukin; Interleukin-2; humanized 3F8 anti-GD2 monoclonal antibody; Carboplatin; Etoposide; Cisplatin; Cyclophosphamide; Doxorubicin; Granulocyte Colony-Stimulating Factor; Filgrastim; Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- R0: COJEC plus G-CSF (Experimental): Patients randomised to G-CSF during induction treatment (Rapid COJEC) received a single daily subcutaneous injection of 5 microgram/kg/day G-CSF (filgrastim) beginning 24 hours after the last chemotherapy dose.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: G-CSF
- R0: COJEC (Active Comparator): Induction treatment (COJEC) without filgrastim Patients randomised to Rapid COJEC alone will receive induction Treatment without G-CSF
  Interventions: Drug: Vincristine; Drug: Carboplatin; Drug: Etoposide; Drug: Cisplatin; Drug: Cyclophosphamide
- R1: BuMel MAT (Active Comparator): The BuMel MAT regimen consists of oral administration of busulphan and the short i.v. infusion of melphalan.
  In July 2007 (amendment 3) oral busulfan was changed to i.v. Busulfan (Busilvex)
  Interventions: Drug: Busulfan; Drug: Melphalan
- R1: CEM MAT (Experimental): The CEM MAT regimen uses three drugs: the dose of Carboplatin must be based on renal function with a target area under the concentration versus time curve (AUC) of 16.4 mg/ml.min, etoposide 350 mg/m2/course and melphalan 210 mg/m2/course
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Melphalan
- R2: ch14.18/CHO (Active Comparator): ch14.18/CHO is given at a dose of 20 mg/m2/day over five days every four weeks for five courses
  Interventions: Drug: ch14.18/CHO
- R2: ch14.18/CHO plus Aldesleukin (Experimental): Patients randomised to receive ch14.18/CHO plus Aldesleukin
  Interventions: Drug: Aldesleukin; Drug: ch14.18/CHO
- R3: COJEC Induction (Active Comparator): Rapid COJEC induction treatment is applied over ten weeks; three different courses are given every ten days:
  Course A (given on days 0 and 40): vincristine, carboplatin, and etoposide Course B (given on days 10, 30, 50, and 70): vincristine and cisplatin Course C (given on days 20 and 60): vincristine, etoposide, and cyclophosphamide
  Interventions: Drug: Vincristine; Drug: Carboplatin; Drug: Etoposide; Drug: Cisplatin; Drug: Cyclophosphamide
- R3: Modified N7 (Experimental): The modified N7 induction is a dose intense induction chemotherapy regimen including two putatively non cross-resistent drug combinations: high-dose cyclophosphamide plus doxorubicin/vincristine (CAV) and high-dose cisplatin/etoposide (P/E).
  Interventions: Drug: Vincristine; Drug: Etoposide; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Doxorubicin
- R4: cnt inf ch14.18/CHO (Active Comparator): ch14.18/CHO is given as continuous Infusion over 10 days at a cumulative dose of 100mg/m2. Patients receive 5 cycles of ch14.18/CHO
  Interventions: Drug: ch14.18/CHO
- R4: cnt inf ch14.18/CHO plus Aldesleukin (Experimental): ch14.18/CHO is given as continuous Infusion over 10 days at a cumulative dose of 100mg/m2. Patients receive 5 cycles of ch14.18/CHO.
  In addition, Aldesleukin is given at a dose of 3 x 10e6 on days 1 to 5 and on days 9, 11, 13, 15, and 17 during ch14.18/CHO infusion
  Interventions: Drug: Aldesleukin; Drug: ch14.18/CHO

INTERVENTIONS:
Drug: Vincristine — given during Rapid COJEC and modified N7 therapy
  Arms: R0: COJEC; R3: COJEC Induction; R3: Modified N7
Drug: Aldesleukin — Aldesleukin is given during MRD Treatment for patients randomised to the arm with IL-2
  Other Names: Interleukin 2, IL-2, IL2
  Arms: R2: ch14.18/CHO plus Aldesleukin; R4: cnt inf ch14.18/CHO plus Aldesleukin
Drug: ch14.18/CHO — ch14.18/CHO antibody is given during MRD treatment
  Other Names: anti GD2 antibody; Dinutuximab beta EUSA; Qarziba®
  Arms: R2: ch14.18/CHO; R2: ch14.18/CHO plus Aldesleukin; R4: cnt inf ch14.18/CHO; R4: cnt inf ch14.18/CHO plus Aldesleukin
Drug: Carboplatin — Carboplatin is given during induction Treatment (R3 randomisation: Rapid COJEC arm)
  Other Names: Paraplatin
  Arms: R0: COJEC; R0: COJEC plus G-CSF; R1: CEM MAT; R3: COJEC Induction
Drug: Etoposide — Etoposide is given during Induction Treatment (both R3 randomisation arms)
  Other Names: VP16
  Arms: R0: COJEC; R0: COJEC plus G-CSF; R1: CEM MAT; R3: COJEC Induction; R3: Modified N7
Drug: Cisplatin — Cisplatin is given during Induction Treatment (both R3 randomisation arms)
  Other Names: CDDP
  Arms: R0: COJEC; R0: COJEC plus G-CSF; R3: COJEC Induction; R3: Modified N7
Drug: Cyclophosphamide — Cyclophosphamid is given during Induction Treatment (both R3 randomisation arms)
  Other Names: Endoxan
  Arms: R0: COJEC; R0: COJEC plus G-CSF; R3: COJEC Induction; R3: Modified N7
Drug: Doxorubicin — Doxorubicin is given during Induction Treatment (R3 arm modified N7)
  Other Names: Adriamycin
  Arms: R3: Modified N7
Drug: G-CSF — G-CSF is given during Induction Treatment
  Other Names: Filgrastim
  Arms: R0: COJEC plus G-CSF
Drug: Busulfan — In case i.v. busulfan is not available, the use of oral busulfan is permitted, although not recommended.
  Other Names: Busilvex; Myleran; Busulphan
  Arms: R1: BuMel MAT
Drug: Melphalan — Melphalan is given during MAT treatment
  Other Names: Alkeran
  Arms: R1: BuMel MAT; R1: CEM MAT

SUMMARY:
This is a randomized study of the European SIOP Neuroblastoma Group (SIOPEN) in high-risk neuroblastoma (stages 2, 3, 4 and 4s MYCN-amplified neuroblastoma, stage 4 MYCN non amplified > 12 months at diagnosis).

The protocol consists of a rapid, dose intensive induction chemotherapy, peripheral blood stem cell harvest, attempted complete excision of the primary tumour, myeloablative therapy followed by peripheral blood stem cell rescue, radiotherapy to the site of the primary tumour and immunotherapy (R4 randomization - isotretinoin and ch14.18/CHO (Dinutuximab beta, Qarziba ®).), with or without s.c. aldesleukin (IL-2)). Patients diagnosed after the closure of R3 randomization will not be R4 randomized. For these patients the use of ch14.18/CHO antibody is recommended without scIL-2 as continuous infusion as standard of care outside of controlled trials. ch14.18/CHO received marketing authorization by EMA in May 2017 (Qarziba ®).

In the induction phase, all patients receive Rapid COJEC following the result of the R3 randomization which was closed on June 8th, 2017 after inclusion of 630 patients as planned.

Following induction treatment peripheral blood stem cell harvest (PBSCH) is performed and complete excision of the primary tumour will be attempted.

Patients with an inadequate metastatic response to allow BuMel MAT followed by PBSCR at the end of induction should receive 2 TVD (Topotecan, Vincristine, Doxorubicin) cycles.

After Rapid COJEC induction, localized patients will proceed to consolidation. Patients aged 12-18 months at diagnosis, with stage 4 neuroblastoma, no MYCN amplification and without segmental chromosomal alterations (SCAs) are thought to have a good prognosis and will stop treatment after induction therapy and surgery to the primary tumour.

Consolidation consists of BuMel MAT based on the results of the R1 randomization followed by peripheral blood stem cell rescue (PBSCR) and radiotherapy to the site of the primary tumour.

The R2 immunotherapy randomization using ch14.18/CHO as 8 hour infusion on 5 consecutive days ( total dose (100mg/m²) with or without aldesleukin (IL-2) alternated with isotretinoin (13-cis-RA) is closed.

The amended R4 immunotherapy randomization using ch14.18/CHO as continuous infusion (total dose 100mg/m² over 10 days) with or without aldesleukin (IL-2) alternated with isotretinoin (13-cis-RA) has accrued according to plan with results pending awaiting data maturity and DMC approval.

DETAILED DESCRIPTION:
In this protocol the term high-risk neuroblastoma refers to children with either

* disseminated disease (INSS stage 4: about 40 to 50% of all neuroblastoma) over the age of one or
* INSS stage 2 and 3 disease with amplification of the MycN proto-oncogene Between 10% and 20% of children with stage 3 and occasional patients with stage 2 disease are characterized by amplification of the MycN gene in their tumours. This biological characteristic has clearly been shown to be associated with a greater risk of relapse and death from disease progression. These patients may benefit from very aggressive treatment and, based on this hypothesis, they are included in this protocol. Infants (< 12 months at diagnosis) with MYCN amplified tumors are included.

Children with this type of presentation and age represent the largest neuroblastoma subgroup. Their prognosis remains poor in most cases and our ability to predict the clinical course and the outcome of the individual patient is modest.

Primary objectives:

R0 randomization: R0 was opened with the study activation in February 2002 and closed in November 2005. The randomized use of G-CSF during COJEC induction resulted in the recommendation of the prophylactic use of G-CSF to prevent episodes of febrile neutropenia (Ladenstein R, Valteau-Couanet D, Brock P, et al. Randomized Trial of prophylactic granulocyte colony-stimulating factor during rapid COJEC induction in pediatric patients with high-risk neuroblastoma: the European HR-NBL1/SIOPEN study. J Clin Oncol. 2010 Jul 20;3516-24).

R1 randomization: R1 was opened with the study activation in February 2002 and closed in 10/2010 following the results showing significant superiority of myeloablative therapy (MAT) with busulfan and melphalan over continuous infusion of carboplatin, etoposide and melphalan (CEM). BuMel is now the standard MAT (Ladenstein R, Pötschger U, Pearson ADJ, et al. Busulfan and melphalan versus carboplatin, etoposide, and melphalan as high-dose chemotherapy for high-risk neuroblastoma (HR-NBL1/SIOPEN): an international, randomized, multi-arm, open-label, phase 3 trial. Lancet Oncol. 2017 Apr;500-14).

R2 randomization: R2 was activated in November 2006 (13-cis retinoic acid +/- chimeric ch14.18/CHO antibody), modified in July 2009 and suspended in August 2013. R2 randomization tested the hypothesis that immunotherapy with ch14.18/CHO and subcutaneous aldesleukin (IL-2, Proleukin®), following MAT and autologous stem cell transplantation, in addition to differentiation therapy with 13-cis retinoic acid, will improve 3-year EFS in patients with high-risk neuroblastoma (ASCO 2016: Ladenstein R, et al J Clin Oncol 34, 2016 (suppl; abstr 10500)).

R3 randomization: R3 was opened in June 2011 and tests the hypothesis that modified N7 induction regimen will improve the metastatic response rates or event free survival (EFS) as compared to Rapid COJEC. As of June 8th, 2017 R3 randomization reached the target of 630 randomized patients as planned. There was no difference in event free survival rate between both regimens (Rapid COJEC and modified N7), but modified N7 had a significantly higher grade 3 and 4 toxicity profile. Therefore, Rapid COJEC is maintained as the SIOPEN standard induction treatment with G-CSF support based on the results of the R0 randomization open from 2002 top 2005 This change has been implemented in amendment 8 of the protocol.

R4 randomization: R4 was activated in April 2014. The SIOPEN long term infusion (LTI) ch14.18/CHO trial successfully lowered the toxicity profile by prolonging the infusion time of the same total ch14.18/CHO antibody dose of 100 mg/m² to 10 days of continuous infusion in relapsed /refractory patients. Hence the HRNBL1/SIOPEN study committee wished to implement this more favorable immunotherapy dosing schedule for the time till the induction question R3 was answered and the HRNBL1/SIOPEN trial may be closed. Considering the high R2 dropout rate of patients unable to receive all immunotherapy cycles in the IL-2 s.c. combination treatment arm and not observing this effect in the current SIOPEN LTI trial, it is suggested to address the IL-2sc dose in the new R4. Therefore the potential synergistic effect of sc IL-2 will be addressed again with 50% of the original s.c. IL-2 dose. The IL-2sc dose will hence be reduced to 3 x 106 IU IL-2/m2/day s.c. in the HR-NBL1/SIOPEN R4 amendment instead of 6 x 106 IU IL-2/m2/day s.c as used in the SIOPEN LTI trial. In the second week of each IT course s.c.IL-2 will be given on days 2, 4, 6, 8, 10 in parallel to the ch14.18/CHO ctn infusion and not during the first 5 days in week 2 as scheduled in the SIOPEN LTI trial. R4 randomization is closed for patients diagnosed after June 8th, 2017, the closure date of R3 randomization. For these patients the use of ch14.18/CHO antibody is recommended without scIL-2 as continuous infusion (total dose 100 mg/m² over 10 days) as standard of care outside of controlled trials without scIL-2. The ch14.18/CHO monoclonal antibody received marketing authorization by EMA in May 2017 (dinutuximab beta, Qarziba®).

ELIGIBILITY:
Inclusion Criteria:

* • Established diagnosis of neuroblastoma according to the International Neuroblastoma Staging System (INSS).

  * Age below 21 years.
  * High risk neuroblastoma defined as either:

    1. INSS stage 2, 3, 4, and 4s with MYCN amplification, or
    2. INSS stage 4 without MYCN amplification aged > 12 months at diagnosis
  * Patients who have received no previous chemotherapy except for one cycle of etoposide and carboplatin (VP16/Carbo). In this situation patients will receive Rapid COJEC induction and the first Rapid COJEC cycle may be replaced by the first cycle VP16/Carbo (etoposide / carboplatin).
  * Written informed consent, including agreement of parents or legal guardian for minors, to enter a randomised study if the criteria for randomisation are met.
  * Tumour cell material available for determination of biological prognostic factors.
  * Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method. Female patients who are lactating must agree to stop breast-feeding.
  * Registration of all eligibility criteria with the data centre within 6 weeks from diagnosis.
  * Provisional follow up of 5 years.
  * National and local ethical committee approval.

Exclusion Criteria:

Any negative answer concerning the inclusion criteria of the study

-

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3300 (Estimated)
Dates: Start 2002-02; Primary Completion 2021-09-30 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (R1: MAT therapy) | Up to three years
  The primary endpoint was the event free survival (EFS) calculated from the date of the first R1 randomisation. The following was considered as event:
  * disease progression or relapse
  * death from any cause
  * second neoplasm
  Patients lost to follow up without event were considered at the date of their last follow up evaluation.
  R1 has been closed in October 2010 following the results of R1 randomisation showing significant superiority for myeloablative therapy (MAT) with busulfan and melphalan (BuMel) in patients with high risk neuroblastoma over MAT with continuous infusion of carboplatin, etoposide and melphalan (CEM). BuMel is now the standard MAT.
Event Free Survival (immunotherapy) | Up to three years
  R2 randomisation comparing immunotherapy with ch14.18/CHO and 13-cis retinoic acid versus 13-cis retinoic acid alone was activated in November 2006. It was amended in July 2009 and compares immunotherapy with anti GD2 antibody ch14.18/CHO with or without aldesleukin (IL-2). Immunotherapy randomisation has been amended in 2014 (R4 randomisation). The ch14.18/CHO antibody is given as continuous Infusion and the randomisation has lasted until the necessary number of patients for R3 randomisation was reached
  The primary endpoint is 3-year event free survival calculated from the date of the second randomisation. The following will be considered as events:
  * disease progression or relapse
  * death from any cause
  * second neoplasm
  Patients lost to follow up without event will be censored at the date of their last follow-up evaluation.
Complete metastatic response (R3: Induction therapy) | Up to 95 days
  R3 randomisation compares two different induction therapy regimen, Rapid COJEC and modified N7.
  Complete metastatic response after induction is defined as:
  * no skeletal uptake on mIBG
  * Negative bone marrow aspirates (by cytomorphology) and trephines
  * Absence of other metastatic sites
Event free survival (R3: Induction therapy) | Up to three years
  R3 randomisation compares two different induction therapy regimen, Rapid COJEC and modified N7.
  The primary endpoint is event free survival calculated from the date of the R3-randomisation. The following will be calculated as events:
  * disease progression or relapse
  * death from any cause
  * second neoplasm
  Patients lost to follow up without event will be censored at the date of their last follow up evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ruth L Ladenstein, MD, MBA, cPM, Principal Investigator — St. Anna Kinderkrebsforschung
Locations (126):
- Australia (6):
  - Women and Children´s Hospital, Adelaide
  - Lady Cilento Children´s Hospital, Brisbane
  - John Hunter Children's Hospital, Newcastle
  - Royal Children's Hospital Melbourne, Parkville
  - Sydney Children's Hospital, Sydney
  - Children´s Hospital Westmead, Westmead
- Austria (5):
  - St. Anna Kinderspital, Vienna, Austra
  - Univ.-Klinik für Kinder- und Jugendheilkunde Graz, Graz
  - Univ.Klinik f. Kinder-u. Jugendheilkunde Innsbruck, Innsbruck
  - Landes- Kinderklinik Linz, Linz
  - St. Johanns Spital LKH Salzburg, Salzburg
- Belgium (6):
  - Cliniques universitaires St-Luc, Brussels
  - Hôpital des Enfants, Brussels
  - University Hospital Gent, Ghent
  - UZ Gasthuisberg, Leuven
  - CHR Citadelle, Liège
  - Clinique de l'Espérance, Montegnée
- University Hospital Motol, Prague, Czechia
- Denmark (4):
  - Aarhus Universitetshospital, Aarhus
  - National State Hospital, Copenhagen
  - University Hospital of Odense, Odense
  - Skejby Hospital, Skejby
- France (13):
  - Hopital d'Enfants Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHR Pellegrin, Le Pellerin
  - Centre Oscar Lambret de Lille, Lille
  - Hopitaux de Marseille La Timone, Marseille
  - CHR de Nantes, Nantes
  - Hôpital Trousseau Paris, Paris
  - Institut Curie, Paris
  - Hôpital American Memorial Hospital, Reims
  - CHU-Saint Etienne, Saint-Etienne
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital D'Enfants de Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif
- Greece (4):
  - "A&P Kyriakou" Children's Hospital, Athens
  - Aghia Sophia Children's Hospital, Athens
  - MITERA Hospital, Heraklion
  - PEPAGNH University Hospital, Heraklion
- Hungary (5):
  - Madarász Children Hospital Budapest, Budapest
  - Semmelweis University of Budapest, Budapest
  - University of Debrecen, Debrecen
  - University of Pecs, Pécs
  - University of Szeged, Szeged
- Dublin: OLHSC, Dublin, Ireland
- Israel (3):
  - Rambam Medical Centre, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - Sheba Medical Center, Tel Aviv
- Italy (22):
  - Ospedale G. Salesi, Ancona
  - Universitŕ degli studi di Bari, Bari
  - Ospedali Riuniti, Bergamo
  - Ospedale S. Orsola, Bologna
  - Ospedale Regionale per le Microcitemie, Cagliari
  - Azienda Ospedaliera di Cosenza, Cosenza
  - Azienda Ospedaliera A. Meyer, Florence
  - Istituto Giannina Gaslini, Genoa
  - Istituto Nazionale Tumori di Milano, Milan
  - Azienda Ospedal. Univ. di Modena, Modena
  - Sec. Univ. degli Studi di Napoli - Policlinico, Napoli
  - Clinica di Oncoematologia Pediatrica Padova, Padua
  - Ospedale dei Bambini, Palermo, Palermo
  - Azienda Ospedaliera Universitaria di Parma-Oncoematologia Pediatrica, Parma
  - Policlinico San Matteo, Pavia
  - Ospedale Civile Spirito Santo, Pescara
  - Ospedale "Infermi ", Rimini
  - Policlinico Borgo Roma, Roma
  - Ospedale Bambino Gesu, Rome
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - O.I.R.M. - S. Anna, Torino
  - Istituto per l'Infanzia "Burlo Garofolo", Trieste
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Rikshospitalet, Oslo
  - University Hospital of North-Norway, Tromsø
- Poland (10):
  - Medical University of Bialystok, Bialystok
  - Medical University of Bydgoszcz, Bydgoszcz
  - Childrens' Hospital in Chorzów, Chorzów
  - Medical University in Gdansk, Gdansk
  - Upper Silesian Centre of Child and Mother's Care, Katowice
  - University Children's Hospital, Krakow
  - Children's University Hospital in Lublin, Lublin
  - University of Medical Sciences Poznan, Poznan
  - Institute Mother and Child, Warsaw
  - Wroclaw Medical University, Wroclaw
- Ipofg-Crl, Lisbon, Portugal
- University Hospital F. D. Roosevelt, Banská Bystrica, Slovakia
- University Children's Hospital Ljubljana, Ljubljana, Slovenia
- Spain (15):
  - H . Materno-Infantil Teresa Herrera, A Coruña
  - H. General de Alicante, Alicante
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Cruces, Bilbao
  - Complejo Hospitalario de Jaen, Jaén
  - H. Monteprincipe, Madrid
  - Hospital 12 de Octubre, Madrid
  - H Central de Asturias, Oviedo
  - H. C. U. de Salamanca, Salamanca
  - H. de Donostia Ntra. Sra. de Aranzazu, San Sebastián
  - H. General de Galicia, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Carlos Haya, Valencia
  - Hospital Infantil La Fe, Valencia
  - H Clinico-Universitario, Zaragoza
- Sweden (2):
  - Queen Silvia's Children's Hospital, Göteburg
  - Childrens Hospital Linkoping, Linköping
- Switzerland (2):
  - University Children's Hospital, Geneva
  - CHUV, Lausanne
- United Kingdom (21):
  - Aberdeen: Royal Aberdeen Children's Hospital, Aberdeen
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrooke's NHS Trust, Cambridge
  - Llandough Hospital, Cardiff
  - Edinburgh Royal Hospital for Sick Children, Edinburgh
  - Glasgow Royal Hospital for Sick Children, Glasgow
  - Leeds: St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Liverpool: Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital, London
  - St Bartholomew's Hospital, London
  - UCLH University College London Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Newcastle: Royal Victoria Infirmary, Newcastle
  - Nottingham: Queen's Medical Centre, Nottingham
  - Oxford: John Radcliffe Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southhampton
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Result] Ladenstein R, Valteau-Couanet D, Brock P, Yaniv I, Castel V, Laureys G, Malis J, Papadakis V, Lacerda A, Ruud E, Kogner P, Garami M, Balwierz W, Schroeder H, Beck-Popovic M, Schreier G, Machin D, Potschger U, Pearson A. Randomized Trial of prophylactic granulocyte colony-stimulating factor during rapid COJEC induction in pediatric patients with high-risk neuroblastoma: the European HR-NBL1/SIOPEN study. J Clin Oncol. 2010 Jul 20;28(21):3516-24. doi: 10.1200/JCO.2009.27.3524. Epub 2010 Jun 21. PMID 20567002
- [Result] Ladenstein R, Potschger U, Pearson ADJ, Brock P, Luksch R, Castel V, Yaniv I, Papadakis V, Laureys G, Malis J, Balwierz W, Ruud E, Kogner P, Schroeder H, de Lacerda AF, Beck-Popovic M, Bician P, Garami M, Trahair T, Canete A, Ambros PF, Holmes K, Gaze M, Schreier G, Garaventa A, Vassal G, Michon J, Valteau-Couanet D; SIOP Europe Neuroblastoma Group (SIOPEN). Busulfan and melphalan versus carboplatin, etoposide, and melphalan as high-dose chemotherapy for high-risk neuroblastoma (HR-NBL1/SIOPEN): an international, randomised, multi-arm, open-label, phase 3 trial. Lancet Oncol. 2017 Apr;18(4):500-514. doi: 10.1016/S1470-2045(17)30070-0. Epub 2017 Mar 2. PMID 28259608
- [Result] Ladenstein R, Potschger U, Valteau-Couanet D, Luksch R, Castel V, Yaniv I, Laureys G, Brock P, Michon JM, Owens C, Trahair T, Chan GCF, Ruud E, Schroeder H, Beck Popovic M, Schreier G, Loibner H, Ambros P, Holmes K, Castellani MR, Gaze MN, Garaventa A, Pearson ADJ, Lode HN. Interleukin 2 with anti-GD2 antibody ch14.18/CHO (dinutuximab beta) in patients with high-risk neuroblastoma (HR-NBL1/SIOPEN): a multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Dec;19(12):1617-1629. doi: 10.1016/S1470-2045(18)30578-3. Epub 2018 Nov 12. PMID 30442501
- [Result] Morgenstern DA, Potschger U, Moreno L, Papadakis V, Owens C, Ash S, Pasqualini C, Luksch R, Garaventa A, Canete A, Elliot M, Wieczorek A, Laureys G, Kogner P, Malis J, Ruud E, Beck-Popovic M, Schleiermacher G, Valteau-Couanet D, Ladenstein R. Risk stratification of high-risk metastatic neuroblastoma: A report from the HR-NBL-1/SIOPEN study. Pediatr Blood Cancer. 2018 Nov;65(11):e27363. doi: 10.1002/pbc.27363. Epub 2018 Jul 17. PMID 30015396
- [Result] Berbegall AP, Bogen D, Potschger U, Beiske K, Bown N, Combaret V, Defferrari R, Jeison M, Mazzocco K, Varesio L, Vicha A, Ash S, Castel V, Coze C, Ladenstein R, Owens C, Papadakis V, Ruud E, Amann G, Sementa AR, Navarro S, Ambros PF, Noguera R, Ambros IM. Heterogeneous MYCN amplification in neuroblastoma: a SIOP Europe Neuroblastoma Study. Br J Cancer. 2018 May;118(11):1502-1512. doi: 10.1038/s41416-018-0098-6. Epub 2018 May 14. PMID 29755120
- [Result] Mueller I, Ehlert K, Endres S, Pill L, Siebert N, Kietz S, Brock P, Garaventa A, Valteau-Couanet D, Janzek E, Hosten N, Zinke A, Barthlen W, Varol E, Loibner H, Ladenstein R, Lode HN. Tolerability, response and outcome of high-risk neuroblastoma patients treated with long-term infusion of anti-GD2 antibody ch14.18/CHO. MAbs. 2018 Jan;10(1):55-61. doi: 10.1080/19420862.2017.1402997. Epub 2017 Dec 5. PMID 29120699
- [Result] Ladenstein R, Potschger U, Valteau-Couanet D, Luksch R, Castel V, Ash S, Laureys G, Brock P, Michon JM, Owens C, Trahair T, Chi Fung Chan G, Ruud E, Schroeder H, Beck-Popovic M, Schreier G, Loibner H, Ambros P, Holmes K, Castellani MR, Gaze MN, Garaventa A, Pearson ADJ, Lode HN. Investigation of the Role of Dinutuximab Beta-Based Immunotherapy in the SIOPEN High-Risk Neuroblastoma 1 Trial (HR-NBL1). Cancers (Basel). 2020 Jan 28;12(2):309. doi: 10.3390/cancers12020309. PMID 32013055
- [Derived] Bellini A, Potschger U, Bernard V, Lapouble E, Baulande S, Ambros PF, Auger N, Beiske K, Bernkopf M, Betts DR, Bhalshankar J, Bown N, de Preter K, Clement N, Combaret V, Font de Mora J, George SL, Jimenez I, Jeison M, Marques B, Martinsson T, Mazzocco K, Morini M, Muhlethaler-Mottet A, Noguera R, Pierron G, Rossing M, Taschner-Mandl S, Van Roy N, Vicha A, Chesler L, Balwierz W, Castel V, Elliott M, Kogner P, Laureys G, Luksch R, Malis J, Popovic-Beck M, Ash S, Delattre O, Valteau-Couanet D, Tweddle DA, Ladenstein R, Schleiermacher G. Frequency and Prognostic Impact of ALK Amplifications and Mutations in the European Neuroblastoma Study Group (SIOPEN) High-Risk Neuroblastoma Trial (HR-NBL1). J Clin Oncol. 2021 Oct 20;39(30):3377-3390. doi: 10.1200/JCO.21.00086. Epub 2021 Jun 11. PMID 34115544
- [Derived] Holmes K, Potschger U, Pearson ADJ, Sarnacki S, Cecchetto G, Gomez-Chacon J, Squire R, Freud E, Bysiek A, Matthyssens LE, Metzelder M, Monclair T, Stenman J, Rygl M, Rasmussen L, Joseph JM, Irtan S, Avanzini S, Godzinski J, Bjornland K, Elliott M, Luksch R, Castel V, Ash S, Balwierz W, Laureys G, Ruud E, Papadakis V, Malis J, Owens C, Schroeder H, Beck-Popovic M, Trahair T, Forjaz de Lacerda A, Ambros PF, Gaze MN, McHugh K, Valteau-Couanet D, Ladenstein RL; International Society of Paediatric Oncology Europe Neuroblastoma Group (SIOPEN). Influence of Surgical Excision on the Survival of Patients With Stage 4 High-Risk Neuroblastoma: A Report From the HR-NBL1/SIOPEN Study. J Clin Oncol. 2020 Sep 1;38(25):2902-2915. doi: 10.1200/JCO.19.03117. Epub 2020 Jul 8. PMID 32639845
- [Derived] Viprey VF, Gregory WM, Corrias MV, Tchirkov A, Swerts K, Vicha A, Dallorso S, Brock P, Luksch R, Valteau-Couanet D, Papadakis V, Laureys G, Pearson AD, Ladenstein R, Burchill SA. Neuroblastoma mRNAs predict outcome in children with stage 4 neuroblastoma: a European HR-NBL1/SIOPEN study. J Clin Oncol. 2014 Apr 1;32(10):1074-83. doi: 10.1200/JCO.2013.53.3604. Epub 2014 Mar 3. PMID 24590653